CLINICAL TRIAL: NCT01483170
Title: Double-blind, Placebo Controlled, Randomized Multiple Ascending Dose Study in Fed Conditions for Ten Days Dosing Regimen With a Loading Dose to Evaluate the Safety, the Tolerability and the Pharmacokinetics of Oral Fexinidazole in 36 Healthy Male Sub-Saharan Volunteers.
Brief Title: Multiple Dose Study to Evaluate Security, Tolerance and Pharmacokinetic of Fexinidazole (Drug Candidate for Human African Trypanosomiasis) Administered With a Loading Dose and With Food
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor tolerability at highest dose
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDiFEX003
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Trypanosomiasis, African
MeSH Terms: conditions — Trypanosomiasis, African | interventions — fexinidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fexinidazole (Experimental)
  Interventions: Drug: Tablets Fexinidazole
- Placebo fexinidazole (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tablets Fexinidazole — Administration of 3 or 4 tablets of 600mg per day during 4 days (loading dose) then administration of 2 tablets of 600mg for 6 days Dosing in fed condition.
  Arms: Fexinidazole
Drug: Placebo — Placebo fexinidazole
  Arms: Placebo fexinidazole

SUMMARY:
This trial will study the tolerability and pharmacokinetic of fexinidazole using two different dosage regimen of repeated administrations. The drug is administered to human healthy volunteers of sub-saharan origin together with food, once a day during 10 days, with a loading dose during 4 days.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives: To assess safety and tolerability of two different fexinidazole dosing regimen, for 10 days repeated administration under fed conditions in healthy male sub-Saharan volunteers.

Secondary objectives: To validate the exposure to fexinidazole, M1 and M2 after different dosing regimens in fed conditions for 10 days in order to evaluate the more appropriate administration regimen for the pivotal phase II/III study.

Methodology/Study Design:

Two dose regimens consisting of repeated oral ascending dose (OAD) dosing in fed condition with two different ascending loading doses for 4 days followed by the same dose for 6 days will be evaluated. The study will be conducted in double-blind conditions for both the clinical and bioanalytical parts.

For each dosing regimen, subjects will reside at the clinical unit from the evening of Day -2 to the afternoon of Day 17 including an 8 days safety follow up (168 h post last dose).

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers 18 to 45 years of age,
* All subjects to be of sub-Saharan African origins with both parents of sub-Saharan African origins too,
* Male subjects with a body mass index (BMI) calculated as weight in kg/(height in m)2 from 18 to 28 kg/m2 inclusive at screening,
* Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study,
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form,
* Light smokers (less than 10 cigarettes per day) or subjects who are non-smokers. No smoking (or use of smoking substitute e.g. nicotine patch) is permitted from screening throughout the study,
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator. These will be measured after resting for 5 min,
* Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV or HCV infection,
* With any clinically significant abnormality following review of pre-study laboratory tests(ASAT, ALAT and alkaline phosphatase (ALP) must be within normal ranges), vital signs, full physical examination and ECG,
* Who are within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health,
* Who forfeit their freedom by administrative or legal award or who were under guardianship,
* Unwilling to give their informed consent,
* Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti-HCV antibodies
* Who have a history of allergy, intolerance or photosensitivity to any drug,
* Who have a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug,
* Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol),
* Who drink more than 8 cups daily of beverage containing caffeine,
* Who have a positive laboratory test for urine drug screening (opiates, cocaine,amphetamine, cannabis, benzodiazepines),
* Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study,
* Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration,
* Who have any clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study,
* Who participated to any clinical trial with an investigational drug in the past 3 months preceding study entry.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Hovsepian, MD, Principal Investigator — SGS Aster
Locations (1):
- SGS Life Sciences, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website — http://www.dndi.org
- See also: Publication combining results of NCT00982904 + NCT01340157 — http://www.dndi.org/wp-content/uploads/2009/06/ClinicalPK_Tarral_FexinidazoleHAT_2014.pdf